CLINICAL TRIAL: NCT02373813
Title: A Randomized Withdrawal Double-blind Study of Etanercept Monotherapy Compared to Methotrexate Monotherapy for Maintenance of Remission in Subjects With Rheumatoid Arthritis
Brief Title: Study of Etanercept Monotherapy vs Methotrexate Monotherapy for Maintenance of Rheumatoid Arthritis Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20110186
Record Dates: First submitted 2015-01-12; First posted 2015-02-27 (Estimated); Results first posted 2020-12-19 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Open Label Run-In: Etanercept plus Methotrexate (Experimental): Etanercept 50 mg weekly by subcutaneous injection plus oral methotrexate 10 to 25 mg weekly for 24 weeks. Participants also receive folic acid as standard of care.
  Interventions: Drug: etanercept pre-filled syringe subcutaneous injection; Drug: Oral methotrexate; Dietary Supplement: Folic acid (non-investigational product)
- Double-Blind Treatment: Methotrexate Monotherapy (Experimental): Oral methotrexate 10 to 25 mg weekly plus placebo for etanercept for 48 weeks. Participants also receive folic acid as standard of care.
  After randomization, a participant experiencing protocol-defined disease worsening will initiate rescue treatment with etanercept 50 mg QW plus methotrexate (10 to 25 mg).
  Interventions: Drug: etanercept pre-filled syringe subcutaneous injection; Drug: Oral methotrexate; Drug: Placebo for etanercept subcutaneous injection; Dietary Supplement: Folic acid (non-investigational product)
- Double-Blind Treatment: Etanercept Monotherapy (Experimental): Etanercept 50 mg weekly by subcutaneous injection plus placebo for methotrexate for 48 weeks. Participants also receive folic acid as standard of care.
  After randomization, a participant experiencing protocol-defined disease worsening will initiate rescue treatment with etanercept 50 mg QW plus methotrexate (10 to 25 mg).
  Interventions: Drug: etanercept pre-filled syringe subcutaneous injection; Drug: Oral methotrexate; Drug: Placebo for methotrexate; Dietary Supplement: Folic acid (non-investigational product)
- Double-Blind Treatment: Etanercept plus Methotrexate (Experimental): Etanercept 50 mg weekly by subcutaneous injection plus oral methotrexate 10 to 25 mg weekly for 48 weeks. Participants also receive folic acid as standard of care.
  After randomization, a participant experiencing protocol-defined disease worsening will continue on the assigned treatments (as rescue treatment).
  Interventions: Drug: etanercept pre-filled syringe subcutaneous injection; Drug: Oral methotrexate; Dietary Supplement: Folic acid (non-investigational product)

INTERVENTIONS:
Drug: etanercept pre-filled syringe subcutaneous injection — etanercept for injection in pre-filled syringes
  Other Names: Enbrel; AMG916
Drug: Oral methotrexate — During the open-label run-in period, methotrexate will be provided as 2.5 mg tablets.
  During the double-blind treatment period, methotrexate will be provided as 2.5 mg capsules.
Drug: Placebo for etanercept subcutaneous injection — etanercept placebo for injection in pre-filled syringes
  Arms: Double-Blind Treatment: Methotrexate Monotherapy
Drug: Placebo for methotrexate — methotrexate placebo capsules
  Arms: Double-Blind Treatment: Etanercept Monotherapy
Dietary Supplement: Folic acid (non-investigational product) — Folic acid 5 to 7 mg per week as per investigator judgment or according to local standard of care.

SUMMARY:
The purpose of this study is to evaluate the efficacy of etanercept monotherapy compared to methotrexate monotherapy on maintenance of remission in participants with rheumatoid arthritis (RA) who were on etanercept plus methotrexate therapy.

This is a multicenter, randomized withdrawal, double-blind controlled study in participants with rheumatoid arthritis on etanercept plus methotrexate therapy who are in very good disease control for 6 months prior to study entry. The study will consist of a 30-day screening period, a 24-week open label run-in period, a 48-week double-blind treatment period and a 30-day safety follow-up period.

ELIGIBILITY:
Inclusion Criteria (Part 1, Run-In Period):

* Subjects must be adults with a history of moderate to severe rheumatoid arthritis;
* Subjects must be in very good rheumatoid arthritis disease control for ≥ 6 months and be in remission as defined by a Simplified Disease Activity Index ≤ 3.3 at screening and at the end of the run-in period.
* Subjects must be on etanercept 50 mg per week plus methotrexate therapy for ≥ 6 months prior to the start of the run-in period. The methotrexate dose must be 10 to 25 mg per week for ≥ 6 months prior to the start of the run-in period and the dose must be stable for ≥ 8 weeks prior to the start of the run-in period.
* Subject has no known history of active tuberculosis, and has a negative test for tuberculosis during screening.

Exclusion Criteria (Part 1, Run-In Period):

* Subject has used biologic disease modifying antirheumatic drug other than etanercept OR has used an oral janus kinase inhibitor ≤ 6 months prior to run-in visit 1
* Subject has any active infection (including chronic or localized infections) for which anti-infectives were indicated within 4 weeks prior to run-in visit 1.
* Subject has known alcohol addiction or dependency or uses alcohol daily.
* Subject has one or more significant concurrent medical conditions per investigator judgment, including the following:

  * poorly controlled diabetes
  * chronic kidney disease stage IIIb, IV, or V
  * symptomatic heart failure (New York Heart Association class II, III, or IV)
  * myocardial infarction or unstable angina pectoris within the past 12 months prior to randomization
  * uncontrolled hypertension
  * severe chronic pulmonary disease (eg, requiring oxygen therapy)
  * multiple sclerosis or any other demyelinating disease
  * major chronic inflammatory disease or connective tissue disease other than rheumatoid arthritis (eg, systemic lupus erythematosus with the exception of secondary Sjögren's syndrome)

Inclusion Criteria (Part 2, Treatment Period):

* SDAI ≤ 3.3 at run-in visit 3
* Subject if female and not at least 2 years postmenopausal or history of hysterectomy, bilateral salpingectomy, or bilateral oophorectomy, has a negative urine pregnancy test at baseline (day 1).

Exclusion Criteria (Part 2, Treatment Period):

* Any clinically significant change in the Part 1 eligibility criteria during the run-in period
* SDAI > 3.3 and ≤ 11 on two consecutive visits at least two weeks apart OR SDAI > 3.3 and ≤ 11 on two or more separate visits OR SDAI > 11 at any time during the run-in period
* Subject has a clinically significant laboratory abnormality during run-in period which in the opinion of the investigator poses a safety risk, will prevent the subject from completing the study, or will interfere with the interpretation of the study results during the run-in period.

NOTE: Other inclusion/exclusion criteria may apply per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (125):
- United States (71):
  - Research Site, Birmingham, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Escondido, California
  - Research Site, Fontana, California
  - Research Site, Hemet, California
  - Research Site, Huntington Beach, California
  - Research Site, La Jolla, California
  - Research Site, Murrieta, California
  - Research Site, Orange, California
  - Research Site, Sacramento, California
  - Research Site, Santa Maria, California
  - Research Site, Torrance, California
  - Research Site, Tustin, California
  - Research Site, Victorville, California
  - Research Site, West Hills, California
  - Research Site, Doral, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Palm Harbor, Florida
  - Research Site, Pensacola, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Meridian, Idaho
  - Research Site, Blue Island, Illinois
  - Research Site, Skokie, Illinois
  - Research Site, Springfield, Illinois
  - Research Site, Granger, Indiana
  - Research Site, Baton Rouge, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Wheaton, Maryland
  - Research Site, Ann Arbor, Michigan
  - Research Site, Detroit, Michigan
  - Research Site, Grand Rapids, Michigan
  - Research Site, Kalamazoo, Michigan
  - Research Site, Lansing, Michigan
  - Research Site, Springfield, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Clifton, New Jersey
  - Research Site, Freehold, New Jersey
  - Research Site, Newark, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Brooklyn, New York
  - Research Site, Great Neck, New York
  - Research Site, New York, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Greenville, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Wynnewood, Pennsylvania
  - Research Site, Wyomissing, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Carrollton, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Cypress, Texas
  - Research Site, League City, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Webster, Texas
  - Research Site, Danville, Virginia
- Research Site, Buenos Aires, Argentina
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (7):
  - Research Site, Winnipeg, Manitoba
  - Research Site, Sydney, Nova Scotia
  - Research Site, Hamilton, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Rimouski, Quebec
  - Research Site, Trois-Rivières, Quebec
- Czechia (2):
  - Research Site, Prague
  - Research Site, Uherské Hradiště
- France (5):
  - Research Site, Bordeaux
  - Research Site, Cahors
  - Research Site, Montpellier
  - Research Site, Orléans
  - Research Site, Paris
- Germany (5):
  - Research Site, Berlin
  - Research Site, Frankfurt am Main
  - Research Site, Hildesheim
  - Research Site, Leipzig
  - Research Site, Püttlingen
- Greece (3):
  - Research Site, Athens
  - Research Site, Heraklion
  - Research Site, Thessaloniki
- Hungary (2):
  - Research Site, Budapest
  - Research Site, Veszprém
- Italy (7):
  - Research Site, Bari
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Napoli
  - Research Site, Reggio Emilia
  - Research Site, Roma
  - Research Site, Verona
- Mexico (4):
  - Research Site, Mexicali, Baja California Norte
  - Research Site, Guadalajara, Jalisco
  - Research Site, Monterrey, Nuevo León
  - Research Site, Chihuahua City
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Karwiany
  - Research Site, Sopot
  - Research Site, Stalowa Wola
- Portugal (3):
  - Research Site, Coimbra
  - Research Site, Lisbon
  - Research Site, Ponte de Lima
- Research Site, Panorama, Western Cape, South Africa
- Spain (8):
  - Research Site, Seville, Andalusia
  - Research Site, Bilbao, Basque Country
  - Research Site, Salamanca, Castille and León
  - Research Site, Barcelona, Catalonia
  - Research Site, A Coruña, Galicia
  - Research Site, Majadahonda, Madrid
  - Research Site, El Palmar, Murcia
  - Research Site, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Curtis JR, Trivedi M, Haraoui B, Emery P, Park GS, Collier DH, Aras GA, Chung J. Defining and characterizing sustained remission in patients with rheumatoid arthritis. Clin Rheumatol. 2018 Apr;37(4):885-893. doi: 10.1007/s10067-017-3923-z. Epub 2017 Dec 9. PMID 29224127
- [Background] Curtis JR, Emery P, Karis E, Haraoui B, Bykerk V, Yen PK, Kricorian G, Chung JB. Etanercept or Methotrexate Withdrawal in Rheumatoid Arthritis Patients in Sustained Remission. Arthritis Rheumatol. 2021 May;73(5):759-768. doi: 10.1002/art.41589. Epub 2021 Mar 24. PMID 33205906
- [Background] Curtis JR, Stolshek B, Emery P, Haraoui B, Karis E, Kricorian G, Collier DH, Yen PK, Bykerk VP. Effects of Disease-Worsening Following Withdrawal of Etanercept or Methotrexate on Patient-Reported Outcomes in Patients With Rheumatoid Arthritis: Results From the SEAM-RA Trial. J Clin Rheumatol. 2023 Jan 1;29(1):16-22. doi: 10.1097/RHU.0000000000001893. Epub 2022 Oct 22. PMID 36459119
- [Derived] Curtis JR, Emery P, Kricorian G, Yen PK, Collier DH, Bykerk V, Haraoui B. Factors Associated With Maintenance of Remission Following Change From Combination Therapy to Monotherapy in Patients With Rheumatoid Arthritis. J Rheumatol. 2023 Sep;50(9):1114-1120. doi: 10.3899/jrheum.2022-1008. Epub 2023 Apr 15. PMID 37061234
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 97 centers in Canada, United States, Argentina, Bulgaria, Czech Republic, Spain, France, Germany, Greece, Hungary, Italy, Mexico, Poland, Portugal, and South Africa. The first participant enrolled on 20 February 2015; the last participant enrolled on 26 June 2018.
Pre-assignment Details: After a 24-week open label run-in period, participants were randomly assigned in a 2:2:1 ratio to one of three treatment groups: methotrexate monotherapy, etanercept monotherapy, or etanercept plus methotrexate.
Groups:
- Double-Blind Treatment: Methotrexate Monotherapy: Oral methotrexate 10 to 25 mg weekly plus placebo for etanercept for 48 weeks. Participants also receive folic acid as standard of care.
  After randomization, a participant experiencing protocol-defined disease worsening initiated rescue treatment with etanercept 50 mg QW plus methotrexate (10 to 25 mg).
- Double-Blind Treatment: Etanercept Monotherapy: Etanercept 50 mg weekly by subcutaneous injection plus placebo to methotrexate for 48 weeks. Participants also receive folic acid as standard of care.
  After randomization, a participant experiencing protocol-defined disease worsening initiated rescue treatment with etanercept 50 mg QW plus methotrexate (10 to 25 mg).
- Double-Blind Treatment: Etanercept Plus Methotrexate: Etanercept 50 mg weekly by subcutaneous injection plus oral methotrexate 10 to 25 mg weekly for 48 weeks. Participants also receive folic acid as standard of care.
  After randomization, a participant experiencing protocol-defined disease worsening continued on the assigned treatments (as rescue treatment).
Period: Run-In Period
Arm/Group | Open Label Run-In: Etanercept Plus Methotrexate | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Started | 371 | 0 | 0 | 0
Treated | 368 | 0 | 0 | 0
Completed | 255 (1 participant who completed the run-in period had no end of study case report form.) | 0 | 0 | 0
Not Completed | 116 | 0 | 0 | 0
Not completed — Other, Not Specified | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 16 | 0 | 0 | 0
Not completed — Decision by Sponsor | 11 | 0 | 0 | 0
Not completed — Protocol Violation | 75 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Not completed — Noncompliance | 1 | 0 | 0 | 0
Not completed — Ineligibility Determined | 3 | 0 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | Open Label Run-In: Etanercept Plus Methotrexate | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Started (One participant who completed the run-in period was not randomized.) | 0 | 101 | 101 | 51
Received Investigational Product (IP) | 0 | 101 | 100 | 51
Received Rescue Treatment | 0 | 52 | 36 | 15
Completed | 0 | 88 | 92 | 47
Not Completed | 0 | 13 | 9 | 4
Not completed — Decision by Sponsor | 0 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 10 | 6 | 3

BASELINE CHARACTERISTICS:
Population: Primary Analysis Set: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate | Total
Number analyzed (Participants) | 101 | 101 | 51 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.4) | 54.8 (12.8) | 55.9 (12.6) | 55.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 77 | 40 | 193
  Male | 25 | 24 | 11 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 19 | 8 | 40
  Not Hispanic or Latino | 88 | 82 | 43 | 213
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 2 | 9
  Asian | 2 | 0 | 1 | 3
  Black | 3 | 7 | 5 | 15
  White | 92 | 86 | 42 | 220
  Other, Not Specified | 0 | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Simplified Disease Activity Index (SDAI) Remission (≤ 3.3) at Week 48: Etanercept Monotherapy vs. Methotrexate Monotherapy
Description: The SDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable, and C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to 86, with higher scores representing worse disease. SDAI remission was defined as a score of ≤ 3.3.
Time Frame: Week 48
Population: Primary Analysis Set: all randomized participants. Nonresponder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy
Number analyzed (Participants) | 101 | 101
percentage of participants | 28.7 | 49.5
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Test type: Superiority; p = 0.004, Chi-squared, Corrected — The risk difference and its p-value were estimated from the chi-squared test with continuity correction; Risk Difference (RD) = 20.8, 95% CI 2-sided [7.6 to 33.9], Standard Error of Mean 6.7

2. Secondary Outcome: Percentage of Participants With SDAI Remission (≤ 3.3) at Week 48: Etanercept and Methotrexate vs. Methotrexate Monotherapy
Description: as for outcome 1
Time Frame: Week 48
Population: Primary Analysis Set: all randomized participants. Nonresponder imputation.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 51
percentage of participants | 28.7 | 52.9
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Test type: Superiority; p = 0.006, Chi-squared, Corrected — The risk difference and its p-value were estimated from the chi-squared test with continuity correction; Risk Difference (RD) = 24.2, 95% CI 2-sided [7.9 to 40.5], Standard Error of Mean 8.3

3. Secondary Outcome: SDAI Score at All Measured Timepoints
Description: The SDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable, and C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to 86, with higher scores representing worse disease.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoints.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Baseline: number analyzed (Participants) | 100 | 101 | 51
  Baseline | 1.29 (0.10) | 1.26 (0.14) | 1.18 (0.17)
  Week 12: number analyzed (Participants) | 100 | 100 | 51
  Week 12 | 7.01 (1.01) | 4.37 (0.75) | 4.39 (1.22)
  Week 24: number analyzed (Participants) | 92 | 96 | 49
  Week 24 | 5.61 (0.98) | 4.98 (0.92) | 3.28 (0.77)
  Week 36: number analyzed (Participants) | 89 | 93 | 48
  Week 36 | 4.03 (0.62) | 2.25 (0.36) | 2.41 (0.40)
  Week 48: number analyzed (Participants) | 84 | 90 | 47
  Week 48 | 3.41 (0.40) | 2.33 (0.23) | 2.86 (0.92)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Baseline; Test type: Superiority; p = 0.58, two sample t-test; Treatment Difference = -0.11, 95% CI 2-sided [-0.48 to 0.27], Standard Error of Mean 0.19
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Baseline; Test type: Superiority; p = 0.85, two sample t-test; Treatment Difference = -0.03, 95% CI 2-sided [-0.37 to 0.31], Standard Error of Mean 0.17
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 12; Test type: Superiority; p = 0.12, two sample t-test; Treatment Difference = -2.61, 95% CI 2-sided [-5.89 to 0.67], Standard Error of Mean 1.66
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 12; Test type: Superiority; p = 0.037, two sample t-test; Treatment Difference = -2.64, 95% CI 2-sided [-5.12 to -0.16], Standard Error of Mean 1.26
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 24; Test type: Superiority; p = 0.063, two sample t-test; Treatment Difference = -2.33, 95% CI 2-sided [-4.80 to 0.13], Standard Error of Mean 1.46
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 24; Test type: Superiority; p = 0.64, two sample t-test; Treatment Difference = -0.63, 95% CI 2-sided [-3.27 to 2.01], Standard Error of Mean 1.34
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 36; Test type: Superiority; p = 0.031, two sample t-test; Treatment Difference = -1.62, 95% CI 2-sided [-3.09 to -0.15], Standard Error of Mean 0.90
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 36; Test type: Superiority; p = 0.015, two sample t-test; Treatment Difference = -1.77, 95% CI 2-sided [-3.20 to -0.35], Standard Error of Mean 0.71
Statistical Analysis 9: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 48; Test type: Superiority; p = 0.58, two sample t-test; Treatment Difference = -0.55, 95% CI 2-sided [-2.55 to 1.45], Standard Error of Mean 0.87
Statistical Analysis 10: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 48; Test type: Superiority; p = 0.020, two sample t-test; Treatment Difference = -1.08, 95% CI 2-sided [-1.99 to -0.17], Standard Error of Mean 0.45

4. Secondary Outcome: Change From Baseline in SDAI Score at All Measured Timepoints
Description: The SDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable, and C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to 86, with higher scores representing worse disease. SDAI remission was defined as a score of ≤ 3.3. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Change at Week 12: number analyzed (Participants) | 99 | 100 | 51
  Change at Week 12 | 5.67 (1.00) | 3.14 (0.75) | 3.21 (1.19)
  Change at Week 24: number analyzed (Participants) | 91 | 96 | 49
  Change at Week 24 | 4.42 (0.98) | 3.78 (0.91) | 2.14 (0.78)
  Change at Week 36: number analyzed (Participants) | 88 | 93 | 48
  Change at Week 36 | 2.90 (0.63) | 1.06 (0.38) | 1.30 (0.43)
  Change at Week 48: number analyzed (Participants) | 83 | 90 | 47
  Change at Week 48 | 2.27 (0.39) | 1.16 (0.24) | 1.77 (0.94)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 12; Test type: Superiority; p = 0.13, two sample t-test; Treatment Difference = -2.46, 95% CI 2-sided [-5.68 to 0.77], Standard Error of Mean 1.63
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 12; Test type: Superiority; p = 0.045, two sample t-test; Treatment Difference = -2.53, 95% CI 2-sided [-4.99 to -0.06], Standard Error of Mean 1.25
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 24; Test type: Superiority; p = 0.071, two sample t-test; Treatment Difference = -2.27, 95% CI 2-sided [-4.75 to 0.20], Standard Error of Mean 1.45
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 24; Test type: Superiority; p = 0.63, two sample t-test; Treatment Difference = -0.64, 95% CI 2-sided [-3.28 to 2.00], Standard Error of Mean 1.34
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 36; Test type: Superiority; p = 0.037, two sample t-test; Treatment Difference = -1.61, 95% CI 2-sided [-3.11 to -0.10], Standard Error of Mean 0.91
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 36; Test type: Superiority; p = 0.013, two sample t-test; Treatment Difference = -1.84, 95% CI 2-sided [-3.30 to -0.39], Standard Error of Mean 0.73
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 48; Test type: Superiority; p = 0.62, two sample t-test; Treatment Difference = -0.51, 95% CI 2-sided [-2.54 to 1.53], Standard Error of Mean 0.88
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 48; Test type: Superiority; p = 0.015, two sample t-test; Treatment Difference = -1.12, 95% CI 2-sided [-2.02 to -0.22], Standard Error of Mean 0.45

5. Secondary Outcome: Disease Activity Score (28 Joint) Calculated Using the Erythrocyte Sedimentation Rate Formula (DAS28-ESR) at All Measured Timepoints
Description: The DAS28-ESR is a modified composite index that was designed to measure disease activity using the number of tender and swollen joints based upon a 28-joint count, ESR in mm/hr, and a 100 mm VAS measuring the participant's general health, from 0 (best) to 100 (worst). DAS28-ESR scores range from 0 to 9.4, where higher scores represent higher disease activity.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Baseline: number analyzed (Participants) | 100 | 100 | 51
  Baseline | 1.80 (0.06) | 1.88 (0.07) | 1.84 (0.09)
  Week 12: number analyzed (Participants) | 99 | 100 | 51
  Week 12 | 2.78 (0.14) | 2.37 (0.12) | 2.32 (0.16)
  Week 24: number analyzed (Participants) | 92 | 95 | 49
  Week 24 | 2.41 (0.13) | 2.54 (0.14) | 2.17 (0.12)
  Week 36: number analyzed (Participants) | 87 | 93 | 48
  Week 36 | 2.32 (0.11) | 2.17 (0.08) | 2.16 (0.12)
  Week 48: number analyzed (Participants) | 85 | 90 | 47
  Week 48 | 2.22 (0.10) | 2.21 (0.08) | 2.11 (0.13)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Baseline; Test type: Superiority; p = 0.75, two sample t-test; Treatment Difference = 0.04, 95% CI 2-sided [-0.19 to 0.26], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Baseline; Test type: Superiority; p = 0.43, two sample t-test; Treatment Difference = 0.08, 95% CI 2-sided [-0.11 to 0.27], Standard Error of Mean 0.10
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 12; Test type: Superiority; p = 0.049, two sample t-test; Treatment Difference = -0.46, 95% CI 2-sided [-0.91 to 0.00], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 12; Test type: Superiority; p = 0.032, two sample t-test; Treatment Difference = -0.40, 95% CI 2-sided [-0.77 to -0.04], Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 24; Test type: Superiority; p = 0.18, two sample t-test; Treatment Difference = -0.24, 95% CI 2-sided [-0.58 to 0.11], Standard Error of Mean 0.20
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 24; Test type: Superiority; p = 0.48, two sample t-test; Treatment Difference = 0.14, 95% CI 2-sided [-0.24 to 0.51], Standard Error of Mean 0.19
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 36; Test type: Superiority; p = 0.35, two sample t-test; Treatment Difference = -0.16, 95% CI 2-sided [-0.51 to 0.18], Standard Error of Mean 0.17
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 36; Test type: Superiority; p = 0.28, two sample t-test; Treatment Difference = -0.15, 95% CI 2-sided [-0.41 to 0.12], Standard Error of Mean 0.13
Statistical Analysis 9: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 48; Test type: Superiority; p = 0.48, two sample t-test; Treatment Difference = -0.12, 95% CI 2-sided [-0.44 to 0.21], Standard Error of Mean 0.16
Statistical Analysis 10: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 48; Test type: Superiority; p = 0.92, two sample t-test; Treatment Difference = -0.01, 95% CI 2-sided [-0.26 to 0.24], Standard Error of Mean 0.13

6. Secondary Outcome: Change From Baseline in DAS28-ESR at All Measured Timepoints
Description: The DAS28-ESR is a modified composite index that was designed to measure disease activity using the number of tender and swollen joints based upon a 28-joint count, ESR in mm/hr, and a 100 mm VAS measuring the participant's general health, from 0 (best) to 100 (worst). DAS28-ESR scores range from 0 to 9.4, where higher scores represent higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Change at Week 12: number analyzed (Participants) | 98 | 100 | 51
  Change at Week 12 | 0.96 (0.13) | 0.50 (0.10) | 0.48 (0.18)
  Change at Week 24: number analyzed (Participants) | 91 | 95 | 49
  Change at Week 24 | 0.65 (0.12) | 0.69 (0.13) | 0.34 (0.11)
  Change at Week 36: number analyzed (Participants) | 86 | 92 | 48
  Change at Week 36 | 0.53 (0.10) | 0.31 (0.08) | 0.35 (0.12)
  Change at Week 48: number analyzed (Participants) | 84 | 89 | 47
  Change at Week 48 | 0.43 (0.09) | 0.34 (0.07) | 0.32 (0.14)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 12; Test type: Superiority; p = 0.032, two sample t-test; Treatment Difference = -0.48, 95% CI 2-sided [-0.91 to -0.04], Standard Error of Mean 0.22
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 12; Test type: Superiority; p = 0.005, two sample t-test; Treatment Difference = -0.46, 95% CI 2-sided [-0.78 to -0.15], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 24; Test type: Superiority; p = 0.058, two sample t-test; Treatment Difference = -0.31, 95% CI 2-sided [-0.63 to 0.01], Standard Error of Mean 0.18
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 24; Test type: Superiority; p = 0.78, two sample t-test; Treatment Difference = 0.05, 95% CI 2-sided [-0.29 to 0.38], Standard Error of Mean 0.17
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 36; Test type: Superiority; p = 0.27, two sample t-test; Treatment Difference = -0.18, 95% CI 2-sided [-0.49 to 0.14], Standard Error of Mean 0.16
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 36; Test type: Superiority; p = 0.078, two sample t-test; Treatment Difference = -0.22, 95% CI 2-sided [-0.47 to 0.03], Standard Error of Mean 0.12
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 48; Test type: Superiority; p = 0.47, two sample t-test; Treatment Difference = -0.12, 95% CI 2-sided [-0.43 to 0.20], Standard Error of Mean 0.16
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 48; Test type: Superiority; p = 0.39, two sample t-test; Treatment Difference = -0.10, 95% CI 2-sided [-0.33 to 0.13], Standard Error of Mean 0.11

7. Secondary Outcome: Disease Activity Score (28 Joint) Using the C-Reactive Protein Formula (DAS28-CRP) at All Measured Timepoints
Description: The DAS28-CRP is a composite index that was designed to measure disease activity using the number of tender and swollen joints based upon a 28-joint count, CRP in mg/L, and a 100 mm VAS measuring the participant's general health from 0 (best) to 100 (worst). DAS28-CRP scores range from 0 to 9.4, where higher scores represent higher disease activity.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given time point.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Baseline: number analyzed (Participants) | 100 | 101 | 51
  Baseline | 1.50 (0.03) | 1.50 (0.04) | 1.54 (0.05)
  Week 12: number analyzed (Participants) | 100 | 100 | 51
  Week 12 | 2.36 (0.13) | 1.91 (0.09) | 1.94 (0.15)
  Week 24: number analyzed (Participants) | 92 | 96 | 49
  Week 24 | 2.15 (0.11) | 2.00 (0.11) | 1.77 (0.09)
  Week 36: number analyzed (Participants) | 89 | 93 | 48
  Week 36 | 1.96 (0.09) | 1.67 (0.06) | 1.72 (0.08)
  Week 48: number analyzed (Participants) | 84 | 90 | 47
  Week 48 | 1.87 (0.07) | 1.67 (0.05) | 1.72 (0.11)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Baseline; Test type: Superiority; p = 0.60, two sample t-test; Treatment Difference = 0.03, 95% CI 2-sided [-0.09 to 0.15], Standard Error of Mean 0.06
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Baseline; Test type: Superiority; p = 0.97, two sample t-test; Treatment Difference = 0.00, 95% CI 2-sided [-0.10 to 0.10], Standard Error of Mean 0.05
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 12; Test type: Superiority; p = 0.044, two sample t-test; Treatment Difference = -0.41, 95% CI 2-sided [-0.82 to -0.01], Standard Error of Mean 0.20
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 12; Test type: Superiority; p = 0.004, two sample t-test; Treatment Difference = -0.45, 95% CI 2-sided [-0.76 to -0.14], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 24; Test type: Superiority; p = 0.009, two sample t-test; Treatment Difference = -0.38, 95% CI 2-sided [-0.66 to -0.10], Standard Error of Mean 0.17
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 24; Test type: Superiority; p = 0.34, two sample t-test; Treatment Difference = -0.15, 95% CI 2-sided [-0.46 to 0.16], Standard Error of Mean 0.16
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 36; Test type: Superiority; p = 0.046, two sample t-test; Treatment Difference = -0.24, 95% CI 2-sided [-0.47 to 0.00], Standard Error of Mean 0.13
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 36; Test type: Superiority; p = 0.006, two sample t-test; Treatment Difference = -0.29, 95% CI 2-sided [-0.49 to -0.08], Standard Error of Mean 0.10
Statistical Analysis 9: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 48; Test type: Superiority; p = 0.25, two sample t-test; Treatment Difference = -0.15, 95% CI 2-sided [-0.40 to -0.10], Standard Error of Mean 0.13
Statistical Analysis 10: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 48; Test type: Superiority; p = 0.021, two sample t-test; Treatment Difference = -0.20, 95% CI 2-sided [-0.37 to -0.03], Standard Error of Mean 0.08

8. Secondary Outcome: Change From Baseline in DAS28-CRP at All Measured Timepoints
Description: The DAS28-CRP is a composite index that was designed to measure disease activity using the number of tender and swollen joints based upon a 28-joint count, CRP in mg/L, and a 100 mm VAS measuring the participant's general health from 0 (best) to 100 (worst). DAS28-CRP scores range from 0 to 9.4, where higher scores represent higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Change at Week 12: number analyzed (Participants) | 99 | 100 | 51
  Change at Week 12 | 0.84 (0.12) | 0.42 (0.09) | 0.41 (0.15)
  Change at Week 24: number analyzed (Participants) | 91 | 96 | 49
  Change at Week 24 | 0.67 (0.11) | 0.52 (0.11) | 0.25 (0.08)
  Change at Week 36: number analyzed (Participants) | 88 | 93 | 48
  Change at Week 36 | 0.49 (0.09) | 0.18 (0.06) | 0.20 (0.08)
  Change at Week 48: number analyzed (Participants) | 83 | 90 | 47
  Change at Week 48 | 0.40 (0.07) | 0.19 (0.04) | 0.21 (0.11)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 12; Test type: Superiority; p = 0.030, two sample t-test; Treatment Difference = -0.43, 95% CI 2-sided [-0.82 to -0.04], Standard Error of Mean 0.20
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 12; Test type: Superiority; p = 0.005, two sample t-test; Treatment Difference = -0.42, 95% CI 2-sided [-0.72 to -0.13], Standard Error of Mean 0.15
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 24; Test type: Superiority; p = 0.002, two sample t-test; Treatment Difference = -0.42, 95% CI 2-sided [-0.69 to -0.15], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 24; Test type: Superiority; p = 0.34, two sample t-test; Treatment Difference = -0.15, 95% CI 2-sided [-0.46 to 0.16], Standard Error of Mean 0.16
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 36; Test type: Superiority; p = 0.014, two sample t-test; Treatment Difference = -0.29, 95% CI 2-sided [-0.52 to -0.06], Standard Error of Mean 0.13
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 36; Test type: Superiority; p = 0.004, two sample t-test; Treatment Difference = -0.30, 95% CI 2-sided [-0.51 to -0.10], Standard Error of Mean 0.10
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 48; Test type: Superiority; p = 0.12, two sample t-test; Treatment Difference = -0.19, 95% CI 2-sided [-0.43 to 0.05], Standard Error of Mean 0.12
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 48; Test type: Superiority; p = 0.010, two sample t-test; Treatment Difference = -0.21, 95% CI 2-sided [-0.37 to -0.05], Standard Error of Mean 0.08

9. Secondary Outcome: Clinical Disease Activity Index (CDAI) at All Measured Timepoints
Description: The CDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, and Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable. The CDAI score ranges from 0 to 76, where a higher score represents worse disease.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Baseline | 1.01 (0.10) | 0.92 (0.13) | 0.71 (0.12)
  Week 12: number analyzed (Participants) | 100 | 101 | 51
  Week 12 | 6.42 (0.98) | 4.08 (0.74) | 3.95 (1.20)
  Week 24: number analyzed (Participants) | 92 | 96 | 49
  Week 24 | 5.07 (0.95) | 4.63 (0.91) | 2.35 (0.60)
  Week 36: number analyzed (Participants) | 89 | 93 | 48
  Week 36 | 3.60 (0.63) | 1.93 (0.36) | 2.04 (0.41)
  Week 48: number analyzed (Participants) | 85 | 92 | 47
  Week 48 | 3.06 (0.38) | 2.00 (0.23) | 2.61 (0.91)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Baseline; Test type: Superiority; p = 0.067, two sample t-test; Treatment Difference = -0.30, 95% CI 2-sided [-0.62 to 0.02], Standard Error of Mean 0.16
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Baseline; Test type: Superiority; p = 0.59, two sample t-test; Treatment Difference = -0.09, 95% CI 2-sided [-0.41 to 0.23], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 12; Test type: Superiority; p = 0.13, two sample t-test; Treatment Difference = -2.46, 95% CI [-5.66 to 0.74], Standard Error of Mean 1.62
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 12; Test type: Superiority; p = 0.059, two sample t-test; Treatment Difference = -2.34, 95% CI 2-sided [-4.76 to 0.09], Standard Error of Mean 1.23
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 24; Test type: Superiority; p = 0.017, two sample t-test; Treatment Difference = -2.72, 95% CI 2-sided [-4.95 to -0.50], Standard Error of Mean 1.38
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 24; Test type: Superiority; p = 0.74, two sample t-test; Treatment Difference = -0.44, 95% CI 2-sided [-3.04 to 2.15], Standard Error of Mean 1.32
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 36; Test type: Superiority; p = 0.039, two sample t-test; Treatment Difference = -1.56, 95% CI 2-sided [-3.03 to -0.08], Standard Error of Mean 0.90
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 36; Test type: Superiority; p = 0.023, two sample t-test; Treatment Difference = -1.66, 95% CI 2-sided [-3.10 to -0.23], Standard Error of Mean 0.72
Statistical Analysis 9: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 48; Test type: Superiority; p = 0.65, two sample t-test; Treatment Difference = -0.46, 95% CI 2-sided [-2.43 to 1.52], Standard Error of Mean 0.85
Statistical Analysis 10: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 48; Test type: Superiority; p = 0.017, two sample t-test; Treatment Difference = -1.07, 95% CI 2-sided [-1.94 to -0.19], Standard Error of Mean 0.44

10. Secondary Outcome: Change From Baseline in CDAI at All Measured Timepoints
Description: The CDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, and Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable. The CDAI score ranges from 0 to 76, where a higher score represents worse disease. A negative change from baseline indicates improvement.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoint.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
score on a scale
  Change at Week 12: number analyzed (Participants) | 100 | 101 | 51
  Change at Week 12 | 5.39 (0.97) | 3.15 (0.73) | 3.24 (1.17)
  Change at Week 24: number analyzed (Participants) | 92 | 96 | 49
  Change at Week 24 | 4.09 (0.95) | 3.75 (0.90) | 1.70 (0.61)
  Change at Week 36: number analyzed (Participants) | 89 | 93 | 48
  Change at Week 36 | 2.69 (0.63) | 1.07 (0.37) | 1.41 (0.40)
  Change at Week 48: number analyzed (Participants) | 85 | 92 | 47
  Change at Week 48 | 2.17 (0.37) | 1.15 (0.23) | 2.00 (0.92)
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 12; Test type: Superiority; p = 0.18, two sample t-test; Treatment Difference = -2.15, 95% CI [-5.29 to 1.00], Standard Error of Mean 1.59
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 12; Test type: Superiority; p = 0.067, two sample t-test; Treatment Difference = -2.24, 95% CI 2-sided [-4.63 to 0.16], Standard Error of Mean 1.21
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 24; Test type: Superiority; p = 0.035, two sample t-test; Treatment Difference = -2.40, 95% CI 2-sided [-4.62 to -0.17], Standard Error of Mean 1.37
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 24; Test type: Superiority; p = 0.79, two sample t-test; Treatment Difference = -0.34, 95% CI 2-sided [-2.91 to 2.23], Standard Error of Mean 1.30
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 36; Test type: Superiority; p = 0.090, two sample t-test; Treatment Difference = -1.27, 95% CI 2-sided [-2.75 to 0.20], Standard Error of Mean 0.91
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 36; Test type: Superiority; p = 0.029, two sample t-test; Treatment Difference = -1.61, 95% CI 2-sided [-3.06 to -0.17], Standard Error of Mean 0.72
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Change at Week 48; Test type: Superiority; p = 0.86, two sample t-test; Treatment Difference = -0.17, 95% CI 2-sided [-2.15 to 1.81], Standard Error of Mean 0.84
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Change at Week 48; Test type: Superiority; p = 0.021, two sample t-test; Treatment Difference = -1.02, 95% CI 2-sided [-1.88 to -0.16], Standard Error of Mean 0.43

11. Secondary Outcome: Percentage of Participants With SDAI Remission (≤ 3.3) at All Measured Timepoints
Description: as for outcome 1
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
percentage of participants
  Baseline: number analyzed (Participants) | 100 | 101 | 51
  Baseline | 96.0 | 92.1 | 96.1
  Week 12: number analyzed (Participants) | 100 | 100 | 51
  Week 12 | 50.0 | 64.0 | 74.5
  Week 24: number analyzed (Participants) | 98 | 99 | 50
  Week 24 | 38.8 | 56.6 | 62.0
  Week 36: number analyzed (Participants) | 97 | 99 | 49
  Week 36 | 36.1 | 55.6 | 55.1
  Week 48: number analyzed (Participants) | 95 | 96 | 48
  Week 48 | 30.5 | 52.1 | 56.3
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Baseline; Test type: Superiority; p = 1.00, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 0.1, 95% CI 2-sided [-6.5 to 6.6], Standard Error of Mean 3.4
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Baseline; Test type: Superiority; p = 0.38, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = -3.9, 95% CI 2-sided [-10.4 to 2.6], Standard Error of Mean 3.3
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 12; Test type: Superiority; p = 0.007, Chi-squared, Corrected; Risk Difference (RD) = 24.5, 95% CI 2-sided [9.0 to 40.0], Standard Error of Mean 7.9
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 12; Test type: Superiority; p = 0.063, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 14.0, 95% CI 2-sided [0.4 to 27.6], Standard Error of Mean 6.9
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 24; Test type: Superiority; p = 0.012, Chi-squared, Corrected; Risk Difference (RD) = 23.2, 95% CI 2-sided [6.7 to 39.8], Standard Error of Mean 8.4
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 24; Test type: Superiority; p = 0.018, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 17.8, 95% CI 2-sided [4.1 to 31.5], Standard Error of Mean 7.0
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 36; Test type: Superiority; p = 0.044, Chi-squared, Corrected; Risk Difference (RD) = 19.0, 95% CI 2-sided [2.1 to 35.9], Standard Error of Mean 8.6
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 36; Test type: Superiority; p = 0.010, Chi-squared, Corrected; Risk Difference (RD) = 19.5, 95% CI 2-sided [5.8 to 33.2], Standard Error of Mean 7.0
Statistical Analysis 9: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 48; Test type: Superiority; p = 0.005, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 25.7, 95% CI 2-sided [8.9 to 42.5], Standard Error of Mean 8.6
Statistical Analysis 10: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 48; Test type: Superiority; p = 0.004, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 21.6, 95% CI 2-sided [7.9 to 35.2], Standard Error of Mean 7.0

12. Secondary Outcome: Percentage of Participants With Boolean Remission at All Measured Timepoints
Description: A participant achieves Boolean remission (66/68-joint count) if all of the following criteria are met at a single timepoint:
  * 68-joint tender joint count ≤ 1
  * 66-joint swollen joint count ≤ 1
  * CRP (mg/dL) ≤ 1
  * Patient's Global Assessment of Disease Activity using a VAS (where 0=no arthritis activity at all and 10=worst arthritis activity imaginable) ≤ 1.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
percentage of participants
  Baseline: number analyzed (Participants) | 100 | 101 | 51
  Baseline | 34.0 | 34.7 | 45.1
  Week 12: number analyzed (Participants) | 100 | 100 | 51
  Week 12 | 18.0 | 23.0 | 19.6
  Week 24: number analyzed (Participants) | 92 | 96 | 49
  Week 24 | 15.2 | 16.7 | 26.5
  Week 36: number analyzed (Participants) | 89 | 93 | 48
  Week 36 | 14.6 | 20.4 | 27.1
  Week 48: number analyzed (Participants) | 84 | 90 | 47
  Week 48 | 20.2 | 13.3 | 25.5
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Baseline; Test type: Superiority; p = 0.25, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 11.1, 95% CI 2-sided [-5.4 to 27.6], Standard Error of Mean 8.4
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Baseline; Test type: Superiority; p = 1.00, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 0.7, 95% CI 2-sided [-12.5 to 13.8], Standard Error of Mean 6.7
Statistical Analysis 3: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 12; Test type: Superiority; p = 0.98, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 1.6, 95% CI 2-sided [-11.6 to 14.9], Standard Error of Mean 6.8
Statistical Analysis 4: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 12; Test type: Superiority; p = 0.48, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 5.0, 95% CI 2-sided [-6.2 to 16.2], Standard Error of Mean 5.7
Statistical Analysis 5: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 24; Test type: Superiority; p = 0.16, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 11.3, 95% CI 2-sided [-3.1 to 25.7], Standard Error of Mean 7.3
Statistical Analysis 6: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 24; Test type: Superiority; p = 0.94, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 1.4, 95% CI 2-sided [-9.0 to 11.9], Standard Error of Mean 5.3
Statistical Analysis 7: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 36; Test type: Superiority; p = 0.12, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 12.5, 95% CI 2-sided [-2.1 to 27.0], Standard Error of Mean 7.4
Statistical Analysis 8: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 36; Test type: Superiority; p = 0.40, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 5.8, 95% CI 2-sided [-5.2 to 16.8], Standard Error of Mean 5.6
Statistical Analysis 9: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Week 48; Test type: Superiority; p = 0.63, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = 5.3, 95% CI 2-sided [-9.8 to 20.4], Standard Error of Mean 7.7
Statistical Analysis 10: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Week 48; Test type: Superiority; p = 0.31, Chi-squared, Corrected — The risk difference and its p-value were estimated from the Chi-squared test with continuity correction; Risk Difference (RD) = -6.9, 95% CI 2-sided [-18.0 to 4.2], Standard Error of Mean 5.7

13. Secondary Outcome: Percentage of Participants With Disease Worsening
Description: Percentage of participants who fulfilled disease-worsening criteria for the first time is presented. Disease worsening is defined as any of the following:
  * an SDAI > 3.3 and ≤ 11 during 2 consecutive visits at least 2 weeks apart
  * SDAI > 3.3 and ≤ 11 on 3 or more separate visits
  * SDAI > 11 after randomization.
  The SDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable, and C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to 86, with higher scores representing worse disease. SDAI remission was defined as a score of ≤ 3.3.
Time Frame: Baseline, Week 12, Week 24, Week 36 and Week 48
Population: Primary Analysis Set: all randomized participants. Observed cases at given timepoint.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 101 | 101 | 51
percentage of participants
  Baseline: number analyzed (Participants) | 100 | 101 | 51
  Baseline | 0.0 | 0.0 | 0.0
  Week 12: number analyzed (Participants) | 100 | 100 | 51
  Week 12 | 42.0 | 23.0 | 17.6
  Week 24: number analyzed (Participants) | 92 | 96 | 49
  Week 24 | 8.7 | 14.6 | 6.1
  Week 36: number analyzed (Participants) | 89 | 93 | 48
  Week 36 | 10.1 | 3.2 | 8.3
  Week 48: number analyzed (Participants) | 84 | 90 | 47
  Week 48 | 4.8 | 0.0 | 4.3

14. Secondary Outcome: Time to Disease Worsening
Description: Disease worsening is defined as any of the following:
  * an SDAI > 3.3 and ≤ 11 during 2 consecutive visits at least 2 weeks apart
  * SDAI > 3.3 and ≤ 11 on 3 or more separate visits
  * SDAI > 11 after randomization.
  The SDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable, and C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to 86, with higher scores representing worse disease. SDAI remission was defined as a score of ≤ 3.3.
Time Frame: up to Week 48
Population: Primary Analysis Set: all randomized participants. Participants with disease worsening.
Measure: Median (Full Range); unit: weeks
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 63 | 40 | 18
weeks | 12.14 [2.3 to 48.7] | 13.21 [3.0 to 36.1] | 18.93 [7.0 to 48.1]
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Test type: Superiority; p < 0.001, Log Rank — P-value was based on the Log-rank test for overall difference on disease-worsening event between two groups
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Test type: Superiority; p < 0.001, Log Rank — P-value was based on the Log-rank test for overall difference on disease-worsening event between two groups

15. Secondary Outcome: Time to Recapture SDAI Remission After Starting Rescue Treatment
Description: In participants who receive rescue treatment during the double-blind treatment period.
  The SDAI is a composite score that is based on the number of tender and swollen joints using a 28-joint count, Physician's Global Assessment of Disease Activity using a visual analog scale (VAS) where 0=no activity at all and 100=worst activity imaginable, Patient's Global Assessment of Disease Activity using a VAS where 0=no arthritis activity at all and 100=worst arthritis activity imaginable, and C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to 86, with higher scores representing worse disease. SDAI remission was defined as a score of ≤ 3.3.
Time Frame: Between rescue and remission or Week 48, whichever comes first.
Population: Rescue Analysis Set: randomized participants who met the definition of disease-worsening and received both at least 1 dose of active rescue therapy etanercept and at least 1 dose of active rescue therapy methotrexate. Participants who recaptured SDAI remission. Observed cases.
Measure: Median (Full Range); unit: weeks
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 37 | 27 | 12
weeks | 11.00 [0.6 to 41.1] | 12.00 [6.0 to 32.0] | 11.36 [6.0 to 35.1]
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Test type: Superiority; p = 0.31, Log Rank — P-value was based on the Log-rank test for overall difference on disease-worsening event between two groups
Statistical Analysis 2: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Monotherapy; Test type: Superiority; p = 0.51, Log Rank — P-value was based on the Log-rank test for overall difference on disease-worsening event between two groups

16. Secondary Outcome: Percentage of Participants Receiving Rescue Treatment Who Experienced SDAI Remission at Week 48
Description: as for outcome 1
Time Frame: Week 48
Population: Rescue Analysis Set: randomized participants who met the definition of disease-worsening and received both at least 1 dose of active rescue therapy etanercept and at least 1 dose of active rescue therapy methotrexate. Observed cases.
Measure: Number; unit: percentage of participants
Arm/Group | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate
Number analyzed (Participants) | 48 | 34 | 15
percentage of participants | 54.2 | 55.9 | 66.7
Statistical Analysis 1: Comparison: Double-Blind Treatment: Methotrexate Monotherapy vs Double-Blind Treatment: Etanercept Plus Methotrexate; Test type: Superiority; p = 0.58, Chi-squared, Corrected; Risk Difference (RD) = 12.5, 95% CI 2-sided [-15.2 to 40.2], Standard Error of Mean 14.1

ADVERSE EVENTS:
Time Frame: Open-Label Run-In period: from enrollment up to 24 weeks. Double-Blind Treatment period: from randomization up to 48 weeks plus 30 days.
Groups:
- Open Label Rescue: Etanercept Plus Methotrexate: After randomization, a participant experiencing protocol-defined disease worsening initiated rescue treatment with etanercept 50 mg QW plus methotrexate (10 to 25 mg).
Arm/Group | Open Label Run-In: Etanercept Plus Methotrexate | Double-Blind Treatment: Methotrexate Monotherapy | Double-Blind Treatment: Etanercept Monotherapy | Double-Blind Treatment: Etanercept Plus Methotrexate | Open Label Rescue: Etanercept Plus Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/368 | 0/100 | 0/99 | 0/53 | 0/103
Serious Adverse Events (participants affected / at risk) | 14/368 | 3/100 | 3/99 | 2/53 | 4/103
Other Adverse Events (participants affected / at risk) | 29/368 | 21/100 | 12/99 | 8/53 | 9/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Run-In: Etanercept Plus Methotrexate (N=368) | Double-Blind Treatment: Methotrexate Monotherapy (N=100) | Double-Blind Treatment: Etanercept Monotherapy (N=99) | Double-Blind Treatment: Etanercept Plus Methotrexate (N=53) | Open Label Rescue: Etanercept Plus Methotrexate (N=103)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abscess intestinal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Abscess of salivary gland (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Run-In: Etanercept Plus Methotrexate (N=368) | Double-Blind Treatment: Methotrexate Monotherapy (N=100) | Double-Blind Treatment: Etanercept Monotherapy (N=99) | Double-Blind Treatment: Etanercept Plus Methotrexate (N=53) | Open Label Rescue: Etanercept Plus Methotrexate (N=103)
Bronchitis (Infections and infestations) | 6 | 0 | 3 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 20 | 3 | 3 | 1 | 7
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 | 18 | 7 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-10-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT02373813/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT02373813/SAP_001.pdf